CLINICAL TRIAL: NCT07249086
Title: Cohort of Nursing Homes (CNH)
Brief Title: Cohort of Nursing Homes
Status: Recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: QTJC2023072
Record Dates: First submitted 2025-08-01; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2024-11

CONDITIONS: Health Status
Keywords: Health status of elderly people; Elderly (people aged 60 or more)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elderly people in medical-nursing care: The elderly people residing in retirement communities with medical facilities
- Elderly people in home care: The elderly people receiving home care

SUMMARY:
The goal of this observational study was to establish cohorts of elderly people in hospital care and elderly people in home care.

DETAILED DESCRIPTION:
This is an observational study that aims to establish a cohort of elderly people through the nursing homes in the area where the "Tianjin Base" is located, and to scientifically observe and measure the changes and improvements in the health of the elderly population brought about by the new medical care model, such as large-scale elderly care complexes, in order to provide a platform for the study of the health of the elderly population, and thus carry out the exploration of a new model of health promotion. Exploration of new models of health promotion. By comparing the elderly care complex with the home health care mode, and exploring the promotion of "active health" awareness of the elderly through intervention, the investigators will explore the appropriate elderly care mode for different conditions of the elderly population, and explore the advantages of the centralized elderly care mode to be promoted to the home elderly population, so as to establish an elderly care mode that is suitable for the elderly population in Tianjin.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participated in this study and provided signed informed consent forms.
* Both male and female.
* Age 60 years old and above.

Exclusion Criteria:

* Unable to participate in physical examinations due to being bedridden or having limited mobility.
* Unable to communicate effectively.
* People cannot participate for other reasons.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly people residing in retirement communities with medical facilities and people receiving home care.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Health status of elderly people | The diseases status of elderly people will be assessed at baseline and at follow-up visits every 3 to 5 years.
  The diseases status of elderly people, including chronic diseases, cancers, and priority diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China